CLINICAL TRIAL: NCT00001733
Title: Screening Study for the Evaluation and Diagnosis of Potential Research Subjects With Retinovascular Diseases
Brief Title: Screening for Studies on Retinovascular Diseases
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980076; 98-EI-0076
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-07-02

CONDITIONS: Diabetic Retinopathy; Macular Degeneration; Pathologic Neovascularization; Retinal Disease
Keywords: Diabetic Retinopathy; Age-Related Macular Degeneration; Neovascularization; Macular Degeneration; Retinal Disease; Diabetes
MeSH Terms: conditions — Diabetic Retinopathy; Macular Degeneration; Neovascularization, Pathologic; Retinal Diseases; Diabetes Mellitus

SUMMARY:
This screening protocol is designed to help recruit patients for National Eye Institute (NEI) studies of the retina, such as diabetic retinopathy and macular degeneration. Patients must meet the specific criteria of a research study, and this protocol serves as a first step for admitting patients to a retinal disease study.

Candidates will undergo a medical history and comprehensive eye examination. The eye examination includes dilation of the pupils to fully examine the retina. In some studies, photographs of the eye are required. This is done using fluorescein angiography. In this procedure, a dye called sodium fluorescein is injected into the blood stream through a vein. After the dye reaches the blood vessels of the eye, photographs are taken of the retina. Other diagnostic procedures may include physical examination, questionnaires, routine laboratory tests and other standard or specialized tests, as needed.

When the screening is completed, patients will be informed of their options to participate in a study. Patients who are ineligible for a current study will be informed of alternative treatments or options. No treatment is offered under this protocol.

DETAILED DESCRIPTION:
This protocol is designed for the screening of patients with presumed retinovascular diseases. It serves as a first step for individuals who may be eligible and wish to participate in National Eye Institute clinical research studies of retinovascular diseases.

Each individual will be thoroughly evaluated during the screening process to determine if they are suitable candidates for inclusion in any of the National Eye Institute ongoing studies. The screening evaluation will include past and current medical histories and an appropriate physical examination, namely a comprehensive eye exam. Other routine diagnostic procedures and tests may also be completed in order to help determine a subject's eligibility. These tests and procedures are of minimal risk and will be described in more detail in section III: "Study Procedures." Once the screening process is completed and their eligibility is assessed, the subjects will be informed of their options to participate in one or more of the current clinical research studies. If no appropriate protocol is identified, recommendations for other treatment options may be given to the individual, their primary doctor, or referring physician.

ELIGIBILITY:
* INCLUSION/EXCLUSION CRITERIA

Inclusion and exclusion criteria vary with the particular protocol for which a patient is being screened.

In addition to those diagnoses currently under study, subjects with unknown conditions that require the establishment of a diagnosis may be eligible for inclusion in this study.

All studies of retinovascular diseases require the subject to have minimum age of 18 years in both men and women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 1998-03-06; Study Completion 2008-07-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States